CLINICAL TRIAL: NCT02936973
Title: Clinical Effect of Catgut Implantation at Acupoints for the Treatment of Simple Obesity: a Multicentre Randomized Controlled Trial
Brief Title: Catgut Implantation at Acupoints for the Treatment of Simple Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei Hospital of Traditional Chinese Medicine (Other)
Collaborators: State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government); Dongzhimen Hospital, Beijing (Other); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201507003; ChiCTR-IOR-16008384 (Registry Identifier: A Multicenter Randomized Controlled Trial of Catgut Implantation at Acupoints for the Treatment of Simple Obesity)
Record Dates: First submitted 2016-10-08; First posted 2016-10-18 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: simple obesity; catgut implantation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real catgut implantation (Experimental): Participants will receive real catgut implantation at acupoints plus lifestyle modification. Participants will receive catgut implantation treatment every two weeks to fulfill a 8-session treatment course.When the acupoints and surrounding skin are disinfected, an absorbable surgical suture of an appropriate length will be embedded into the muscular layer or subcutaneous tissue of the acupoints by the specified disposable embedding needles. The absorbable surgical suture then stimulated those points over a long period.
  Interventions: Device: Real catgut implantation at acupoints
- sham catgut implantation (Sham Comparator): Participants will receive sham catgut implantation at acupoints and lifestyle modification every two weeks to fulfill a 8-session treatment course.The operation process will be similar to that applied in the real catgut implantation group. Empty needles without catgut will be pushed into the chosen position, to a depth equivalent to that used for catgut implantation at acupoints. The frequency and duration were the the same as the catgut embedding group.
  Interventions: Device: sham catgut implantation at acupoints

INTERVENTIONS:
Device: Real catgut implantation at acupoints — 1. Absorbable surgical suture will be embedded in acupoints as below. Group A ：Zhigou (TE 6), Tianshu (ST25), Weishu (BL21), Zhongwan (CV12) and Zusanli (ST36); Group B ：Quchi (LI11), Huaroumen (ST24), Pishu (BL20), Shuifen (CV9), and Fenglong (ST40). Each group will be used alternatively and treated once every 2 weeks.
  2. lifestyle intervention :Experienced nutritionists calculated every participant's basal metabolic rate,then designed a proper diet and exercise treatment for them. During the treatment, a diet and exercise diary will be distributed to the patients, and detailed guidance concerning their diet and exercise will be provided according to the diary. The patients should be encouraged to maintain the diet and exercise diary for at least 4 days per week .
  Arms: Real catgut implantation
Device: sham catgut implantation at acupoints — Empty needles without catgut will be pushed into the chosen position as below :Group A ：1 cun lateral from the Zhigou (TE 6), Tianshu (ST25), Weishu (BL21), Zhongwan (CV12) and Zusanli (ST36); Group B ：1 cun lateral from the Quchi (LI11), Huaroumen (ST24), Pishu (BL20), Shuifen (CV9), and Fenglong (ST40).Those two groups of acupoints will ultimately be selected for alternative treatment. Each group will be used alternatively and treated once every 2 weeks.
  lifestyle intervention :It will be performed as the same as the real catgut implantation at acupoints group.
  Arms: sham catgut implantation

SUMMARY:
The primary objective of this multicenter randomized controlled trial is to evaluate treatment effectiveness of intervening simple obesity people with catgut implantation at preferred acupoints, which excludes placebo effect; the secondary objective is to evaluate safety and superiority of treating simple obesity with catgut implantation at acupoints to provide high-level evidence for it clinically.

DETAILED DESCRIPTION:
This randomized, double-blind sham-controlled clinical trial will be conducted at Hubei Provincial Hospital of TCM, Dongzhimen Hospital Beijing University of Chinese Medicine and the First Hospital of Hunan University of Chinese Medicine. This study includes the following time points: a treatment period of 16 weeks after screening and a follow-up period of 24 weeks. The total study period will be 40 weeks. All patients will be randomized into the real catgut implantation at acupoints group or the sham catgut implantation at acupoints group.The primary outcome measurement of this study is the rate of waistline reduction compared with baseline. The secondary outcome measurements are the rate of reduction of weight, BMI, hipline, WHR and PBF, and changes in the IWQOL-Lite compared with baseline. These parameters will be evaluated at week 0, week 4, week 8, week 12, week 16, week 28 and week 40. Changes in SF-36, HAD and SES compared with baseline will be evaluated at week 0, week 16 and week 40. SF-36 and IWQOL-Lite will be used to evaluate obese patient quality of life. HAD and SES will be used to evaluate psychological status. In addition, hepatorenal function, blood fat, liver bladder spleen colour ultrasound, FBG and insulin concentration will be used to evaluate whether catgut implantation at acupoints can improve the physiological function of obese patients.

ELIGIBILITY:
Inclusion criteria

Patients recruited for this study should meet the following inclusion criteria:

1. meeting the diagnosis standard for simple obesity in Redefinition and Processing of Obesity in Asia & Pacific Area released by WHO in February 2000;
2. age: 18-45;
3. BMI: 25≤BMI<30;
4. waistline: males ≥95 cm; females ≥85 cm;
5. smokers have not changed their smoking habits for at least 2 months;
6. willing to accept the above-described intervention methods.

Exclusion criteria

Patients with any of the following criteria will be excluded from the study:

1. endocrine disease (such as polycystic ovarian syndrome, Cushing's Disease, and hypothyroidism, among others);
2. gestational diabetes or uncontrolled hypertension (SBP ≥160 mmHg; DBP ≥100 mmHg) [23], or lung, heart, liver or kidney disease;
3. nervous system disease or mental disorders, history of hospitalized depression, two instances of paralepsy or suicidal tendency;
4. history of clinical diagnosis of an eating disorder , such as bulimia or cynorexia, anorexia; or weight changes greater than 5 kg in the previous 3 months;
5. history of weight loss with surgery or a history of post-operative adhesion;
6. having taken drugs with a known influence on weight or appetite in the previous 3 months, such as diet pills, corticosteroid drugs, anti-depression drugs, diazepam drugs, nonselective body antihistamine, nicotine replacements, or hypoglycaemic drugs, or planning to give up smoking and drinking;
7. pregnancy, lactation, or planning to become pregnant within 40 weeks;
8. received catgut implantation at acupoints;
9. participated in clinical research on obesity in the previous 3 months ;
10. protein allergy and scars;
11. skin disease such as eczema and psoriasis;
12. coagulation disorders, taking warfarin, heparin or other anticoagulant drugs;
13. not cooperative or cannot maintain treatment during the study period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
the rate of waistline reduction compared with baseline | week4 ,week8,week12,week16,week28,week40.

SECONDARY OUTCOMES:
the rate of reduction of weight compared with baseline | week4 ,week8,week12,week16,week28,week40.
the rate of reduction of body mass index compared with baseline | week4 ,week8,week12,week16,week28,week40.
the rate of reduction of hipline compared with baseline | week4 ,week8,week12,week16,week28,week40.
the rate of reduction of waist-hip ratio compared with baseline | week4 ,week8,week12,week16,week28,week40.
the rate of reduction of percentage of body fat compared with baseline | week4 ,week8,week12,week16,week28,week40.
changes in IWQOL - Lite scale score compared with baseline | week4 ,week8,week12,week16,week28,week40.
changes in SF - 36 life quality scale score compared with baseline | week4 ,week16,week40.
changes in HAD scale score compared with baseline | week4 ,week16,week40.
changes in self-esteem scale score compared with baseline | week4 ,week16,week40.
changes in serum total cholesterol compared with baseline | week16.
changes in serum triglyceride compared with baseline | week16.
changes in low-density lipoprotein cholesterol (LDL-C) compared with baseline | week16.
changes in High-density lipoprotein cholesterol(HDL-C) compared with baseline | week16.
changes in fasting blood-glucose （FBG）compared with baseline | week16.
changes in fasting insulin ( FINS) compared with baseline | week16.
The adverse effects of catgut implantation at acupoints and as measured by number of participants with adverse events. | from week 2 to week 16.
  The adverse effects of catgut implantation at acupoints include local swelling, pruritus, fever, festering and unbearable pain. In the event of an adverse effect during the trial, the patient should immediately contact the physician. All adverse effects should be promptly recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongyu Zhou, Professor, Principal Investigator — Hubei Hospital of Traditional Chinese Medicine
Locations (1):
- Hubei Provincial Hospital of Traditional Chinese Medicine, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
the data will be published in the form of public papers before May 2019 for public inquiries

REFERENCES:
- [Background] Scheen AJ, Finer N, Hollander P, Jensen MD, Van Gaal LF, RIO-Diabetes Study Group. Efficacy and tolerability of rimonabant in overweight or obese patients with type 2 diabetes: a randomised controlled study. Lancet. 2006;368:1660-72. Preljevic VT, Østhus TB, Sandvik L, Opjordsmoen S, Nordhus IH, Os I, et al. Screening for anxiety and depression in dialysis patients: comparison of the Hospital Anxiety and Depression Scale and the Beck Depression Inventory. J Psychosom Res. 2012;73:139-44. Van Gaal LF, Rissanen AM, Scheen AJ, Ziegler O, Rössner S, RIO-Europe Study Group. Effects of the cannabinoid-1 receptor blocker rimonabant onweight reduction and cardiovascular risk factors in overweight patients: 1-year experience from the RIO-Europe study. Lancet. 2005;365:1389-97. Rosenberg M. Society and the adolescent self-image. Princeton, NJ: Princeton University Press; 1965. World Health Organization, Regional Office for the Western Pacific. The Asia-Pacific perspective: redefining obesity and its treatment. Sydney: Health Communications Australia; 2000. Astrup A, Madsbad S, Breum L, Jensen TJ, Kroustrup JP, Larsen TM. Effect of tesofensine on bodyweight loss, body composition, and quality of life in obese patients: a randomised, double-blind, placebo-controlled trial. Lancet. 2008;372:1906-13. MacPherson H, White A, Cummings M, Jobst KA, Rose K, Niemtzow RC, et al. Standards for reporting interventions in controlled trials of acupuncture: the STRICTA recommendations. J Altern Complement Med. 2002;8:85 - 9. Ralph JL, Von Ah D, Scheett AJ, Hoverson BS, Anderson CM. Diet assessment methods: a guide for oncology nurses. Clin J Oncol Nurs. 2011;15:E114 - 21. James WP, Astrup A, Finer N, Hilsted J, Kopelman P, Rössner S, et al. Effect of sibutramine on weight maintenance after weight loss: a randomised trial. STORM Study Group. Sibutramine Trial of Obesity Reduction and Maintenance Lancet. 2000;356:2119-25.
- [Derived] Chen X, Huang W, Wei D, Zhao JP, Zhang W, Ding DG, Jiao Y, Pan HL, Zhang JJ, Zhong F, Gao F, Jin YT, Zheng YW, Zhang YJ, Huang Q, Zeng XT, Zhou ZY. Effect of Acupoint Catgut Embedding for Middle-Aged Obesity: A Multicentre, Randomised, Sham-Controlled Trial. Evid Based Complement Alternat Med. 2022 Feb 27;2022:4780019. doi: 10.1155/2022/4780019. eCollection 2022. PMID 35265146
- [Derived] Chen X, Huang W, Wei D, Ding DG, Jiao Y, Pan HL, Jin YT, Zheng YW, Zhang YJ, Zhang YR, Liu YR, Zhou ZY. Clinical effect of catgut implantation at acupoints for the treatment of simple obesity: A multicentre randomized controlled trial. Medicine (Baltimore). 2020 Nov 25;99(48):e23390. doi: 10.1097/MD.0000000000023390. PMID 33235115
- See also: Related Info — http://online.liebertpub.com/doi/abs/10.1089/107555302753507212
- See also: Related Info — https://cjon.ons.org/cjon/15/6/diet-assessment-methods
- See also: Related Info — http://www.thelancet.com/journals/lancet/article/PIIS0140-6736(00)03491-7/abstract